CLINICAL TRIAL: NCT03744611
Title: Efficacy and Safety of Cortex Eucommiae (CE: Eucommia Ulmoides Oliver Extract) in Subjects With Mild Osteoarthritis: a 12-week, Multi-center, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Cortex Eucommiae (CE: Eucommia Ulmoides Oliver Extract) in Subjects With Mild Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JS-CT-2018-05
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis
Keywords: Cortex Eucommiae; mild OA
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortex Eucommiae(CE) (Experimental): CE capsule administered orally twice daily for 12 weeks.
  Interventions: Dietary Supplement: CE
- Placebo (Placebo Comparator): Placebo capsule administered orally twice daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CE — 550mg capsule (Eucommia ulmoides Oliver extract)
  Arms: Cortex Eucommiae(CE)
Dietary Supplement: Placebo — 550mg capsule (Placebo)
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Cortex Eucommiae (CE: Eucommia ulmoides Oliver extract) in subjects with mild osteoarthritis (OA).

DETAILED DESCRIPTION:
This is a 12-week, multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of Cortex Eucommiae (CE: Eucommia ulmoides Oliver extract) in subjects with mild OA. One hundred subjects with mild OA will be recruited and randomly divided into 2 groups, each group will receive Cortex Eucommiae (CE: Eucommia ulmoides Oliver extract) or placebo and will take CE or placebo for 12 weeks. Outcomes will be evaluated by self-administered questionnaires and lab test results. The hypothesis is that Cortex Eucommiae (CE: Eucommia ulmoides Oliver extract) which as a dietary supplementation may slow down or reverse OA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 40 ~ 75 years of age
* VAS (Visual Analogue Scale) over 30mm
* Kellgren & Lawrence Grade I~II by X-ray
* Subject who agrees to participate in this clinical trial by themselves and signs the Informed Consent Form (ICF)

Exclusion Criteria:

* Joint space under 2mm by X-ray
* Kellgren & Lawrence Grade over III with osteophyte, irregularly-shaped auricular surfaces, or subchondral bone cyst by X-ray
* Subjects who diagnosed inflammatory arthritis (rheumatoid arthritis, fibromyalgia, systemic lupus erythematosus, septic arthtritis, gout), or articulation fracture with abnormal values at ESR and CRP
* Subjects who diagnosed cardiovascular disease, immune disease, infectious diseases, tumor diseases
* Subjects having gastrointestinal diseases
* Uncontrolled hypertension patients (Blood pressure ≥ 160/100mmHg)
* Uncontrolled diabetes melitusl patients (fasting glucose level ≥ 180mg/dl)
* Subjects have attended abnormal values at AST or ALT (3 times excess at upper limit of the normal values)
* Subjects have attended abnormal values at creatinine (2 times excess at upper limit of the normal values)
* Pregnancy, breast-feeding, or subjects who have a plan to pregnancy within 3 months
* Use of osteoarthritis treatment drugs or dietary supplements within 2 weeks prior to screening
* History of osteoarthritis treatment therapy within 2 weeks prior to screening
* Psychiatric disorder patient (schizophrenia, depressive disorder, drug abuse)
* Have participated in another clinical trial within the 3 months prior to screening
* Subjects who have hypersensitivity history about investigational product
* Have difficulty to be participated in this clinical trial by investigator's decision

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale) | Change of the week 6, 12 from baseline
  VAS to measure changes in joint pain on 6, 12 weeks after administration in comparison with baseline
K-WOMAC (Korean-Western Ontario and McMaster Universities) | Change of the week 6, 12 from baseline
  K-WOMAC to measure changes in joint pain and function on 6, 12 weeks after administration in comparison with baseline
KSF-36 (Korean-Short Form Health Survey 36) | Change of the week 6, 12 from baseline
  KSF-36 to measure changes in physical and mental function on 6, 12 weeks after administration in comparison with baseline

SECONDARY OUTCOMES:
Subject's global impression of change scale | 6 weeks, 12 weeks
  The change in activity limitations, symptoms, emotions and overall quality of life, related to painful condition that is assessed by subject
  Level of Quality
  * Excellent: substantial overall improvement of symptoms
  * Good: overall improvement of symptoms
  * Neutral: no change compared with before
  * Worse: overall deterioration of symptoms
  * Very much worse: substantial overall deterioration of symptoms
Investigator's global impression of change scale | 6 weeks, 12 weeks
  The change in activity limitations, symptoms, emotions and overall quality of life, related to painful condition that is assessed by investigator
  Level of Quality
  * Excellent: substantial overall improvement of symptoms
  * Good: overall improvement of symptoms
  * Neutral: no change compared with before
  * Worse: overall deterioration of symptoms
  * Very much worse: substantial overall deterioration of symptoms
ESR (Erythrocyte sedimentation rate) | Change of the week 12 from baseline
  ESR to measure changes in blood inflammatory marker on 12 weeks after administration in comparison with baseline
CRP (C-reactive protein) | Change of the week 12 from baseline
  CRP to measure changes in blood inflammatory marker on 12 weeks after administration in comparison with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Yeong Ahn, PhD, Study Director — Jaseng Medical Foundation; Jae-Heung Cho, KMD,PhD, Principal Investigator — Kyung Hee University at Gangdong; Dongwoo Nam, KMD,PhD, Principal Investigator — Kyunghee University; Eun-Jung Kim, KMD,PhD, Principal Investigator — DongGuk University; In-Hyuk Ha, KMD,PhD, Study Chair — Jaseng Medical Foundation
Locations (3):
- South Korea (3):
  - Kyung Hee University Korean Medicine Hospital, Seoul
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul
  - Dongguk University Bundang Oriental Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahn HY, Cho JH, Nam D, Kim EJ, Ha IH. Efficacy and safety of Cortex Eucommiae (Eucommia ulmoides Oliver) extract in subjects with mild osteoarthritis: Study protocol for a 12-week, multicenter, randomized, double-blind, placebo-controlled trial. Medicine (Baltimore). 2019 Dec;98(50):e18318. doi: 10.1097/MD.0000000000018318. PMID 31852118